CLINICAL TRIAL: NCT05544812
Title: The First Affilcated Hosipital ,the Air Force Medical University
Brief Title: A Small-sample, Real-world Study of Sintilimab Plus Bevacizumab/Cetuximab Plus XELOX Regimen for Conversion Therapy in Patients With Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: yangjianjun-2
Record Dates: First submitted 2022-09-02; First posted 2022-09-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental: Patients in this group had previously received the following treatment regimens:
  Oxaliplatin :130 mg/m2, D1, Q3W; Capecitabine :1000mg/m2, bid q2w Sintilimab for injection :200mg, D1, Q3W Bevacizumab :7.5mg/kg, D1, Q3W or cetuximab :500 mg/m, D1, Q2W
  Interventions: Drug: Sintilimab ，bevcizumab/cetuximab，XELOX

INTERVENTIONS:
Drug: Sintilimab ，bevcizumab/cetuximab，XELOX — Patients in this group had previously received the following treatment regimens:
  Oxaliplatin :130 mg/m2, D1, Q3W; Capecitabine :1000mg/m2, bid q2w Sintilimab for injection :200mg, D1, Q3W Bevacizumab :7.5mg/kg, D1, Q3W or cetuximab :500 mg/m, D1, Q2W

SUMMARY:
The purpose of this study is to acssess the efficacy and the safety of Sintilimab plus bevacizumab/cetuximab plus XELOX regimen for conversion therapy in patients with advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients had to meet all the following conditions to be enrolled in this study:

Pathological diagnosis of colorectal adenocarcinoma; Ambulatory cases, aged 18-75 years; ECOG score less than or equal to 1; Have not received anti-tumor therapy (such as surgery, radiotherapy, chemotherapy, targeted therapy, immunological therapy);

Baseline blood routine and biochemical parameters of the subjects met the following criteria:

1. Blood routine examination standards shall meet: A. WBC & GT; 4.0 x 10 / L; b. ANC > 1.5 x 10 / L; C. the ANC acuity 1.5 x 109 / L; D. HB ≥ 80 g/L; E. PLT acuity 100 x 109 / L;
2. Biochemical tests shall meet the following standards:

A. TBIL 1.5 x ULN or less; B. ALT and AST & LT; 2.5×ULN, ALT and AST & LT for patients with liver metastases; 5 x ULN; C. BUN and Cr ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50 mL/min(Cockcroft-Gault formula).

No history of other tumors； Be willing and able to follow the protocol during the study； Withdraw from the study at any time during the study without any loss; No history of other tumors; Be willing and able to follow the protocol during the study; Written informed consent was provided prior to study screening and was understood by the patient； Expected life ≥ 6 months

Exclusion Criteria:

-

Patients were not admitted to the study if they met any of the following criteria:

1. Cured basal cell carcinoma of the skin and uterus in patients with other malignancies in the past； Cervical carcinoma in situ is excluded;
2. Patients with known positive HER-2 test;
3. Pregnant or lactating women are in the reproductive period and have not taken effective contraceptive measures, or have fertility requirements during the study period;
4. Serious and uncontrolled medical diseases and infections; Chronic bowel disease or short bowel syndrome;
5. Major organ failure, such as compensatory cardiopulmonary, liver and kidney failure; Severe abnormal liver and kidney function metabolism, affecting the normal drug metabolism;
6. Patients with investigator-identified propensity for gastrointestinal bleeding and/or abnormal coagulation (INR & GT; 1.5);
7. Active HBV or HCV;
8. Patients with peripheral neuropathy NCT-CTCAE ≥ grade 2;
9. Patients who were allergic to the drug in the study protocol were not suitable to participate in the clinical study.
10. Patients with rheumatic diseases, such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, such as ankylosing spondylitis, psoriasis arthritis, gout, pseudogout, etc. Laboratory tests included positive antinuclear antibody, anti-DS-DNA antibody, anti-SM antibody, anti-phospholipid antibody, HLA-B27, rheumatoid factor (RF-igm), anti-cyclic citrulline (CCP) antibody, rheumatoid factor IgG and IgA, antinuclear factor, anti-keratin antibody, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with initially unresectable advanced colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
AE | 2-year
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V5.0

SECONDARY OUTCOMES:
ORR | 1-year
  Objective response rate (ORR): Defined as the proportion of patients who achieved a prespecified reduction in tumor volume and maintained a minimum duration, including cases with CR and PR. Objective tumor response was assessed by an independent review committee using the Response Assessment Criteria for solid Tumors (RECIST 1.1 criteria).
DCR | 1-year
  The proportion of all subjects who were randomized and whose best overall response (BOR) was complete response (CR), partial response (PR), and stable disease (SD) according to RECIST1.1 criteria.
OS | 2-year
  It was defined as the time between the start of randomization and the death of the subject from any cause and was calculated in the intention-to-treat population (ITT).

CONTACTS AND LOCATIONS:
Locations (1):
- Yang Jianjun, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No